CLINICAL TRIAL: NCT05879874
Title: Prospective Evaluation of Neurofilament Light Chains as a Biomarker in Hereditary Amyloidosis (ATTRv), Including Correlation With Various Measurements of Disease Severity and Progression.
Brief Title: Prospective Evaluation of NfL as a Biomarker in ATTRv
Acronym: NfLInATTRv
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID5545
Record Dates: First submitted 2023-05-09; First posted 2023-05-30 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Amyloidosis, Hereditary
Keywords: ATTRv; NfL; Disease progression; Disease severity
MeSH Terms: conditions — Amyloidosis, Familial; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ATTR amyloidosis is a rare and progressively disabling disease caused by the deposition of misfolded TTR protein in multiple tissues including the nerves, heart, and gastrointestinal tract. Polyneuropathy (PN) and cardiomyopathy (CM) are the two most frequent phenotypes and many patients presented a mixed picture of PN and CM. There are different methods to search for the existence and extent of PN and disability caused by ATTR amyloidosis (e.g. mNIS+7, Norfol, QoL-DN), these methods may not be sensitive enough to search for the onset of disease in patients carrying the pathogenic TTR variants or progression of PN in patients undergoing treatment. Also, some of the available methods can be difficult and time-consuming to perform. For this reason, there is a need for sensitive biomarkers that can aid in the investigation and follow-up of PN in patients with hATTR amyloidosis. NfL, a well-known biomarker of nerve damage due to both central and peripheral nervous system disorders, was recently evaluated as a potential biomarker of nerve damage in patients with hATTR amyloidosis. The results of this study can help understand the potential value of NfL in patients with PN of hATTR amyloidosis establishing i changes levels of this biomarker in response to different pathology-specific treatment options correlation between NfL levels and different ratings clinics. The primary objective of the study is to establish the potential of NfL as a biomarker of severity of polyneuropathy, progression and response to treatment in patients with symptomatic hATTR amyloidosis.

DETAILED DESCRIPTION:
INTRODUCTION, BACKGROUND AND RATIONALE ATTR amyloidosis is a rare and progressively disabling disorder caused by the deposition of the misfolded TTR protein in multiple tissues including nerves, heart and gastro-intestinal tract. The disease can be caused by a misfolded or wild type variant of the TTR protein. Polyneuropathy (PN) and cardiomyopathy (CM) are the two most frequent phenotypes, and many patients have a mixed picture of PN and CM.

There are different methods to research the existence and extent of PN and the disability caused by ATTR amyloidosis (e.g. mNIS+7, Norfol, QoL-DN), these methods may not be sensitive enough to search for disease onset in patients carrying pathogenic TTR variants or PN progression in patients undergoing treatment. In addition, some of the available methods can be difficult and time-consuming. For this reason, there is a need for sensitive biomarkers that can aid in PN research and follow-up in patients with hATTR amyloidosis.

NfL, a well-known biomarker of nerve damage due to both central and peripheral nervous system disorders, has recently been evaluated as a potential biomarker of nerve damage in patients with hATTR amyloidosis.

The results of this study may contribute to understanding the potential value of NfL in patients with hATTR amyloidosis PN by establishing changes in levels of this biomarker in response to different disease-specific treatment options and the correlation between NfL levels and different clinical assessments.

OBJECTIVES

Primary Objective The primary objective of the study is to establish the potential of NfL as a biomarker of severity of polyneuropathy, progression and response to treatment in patients with symptomatic hATTR amyloidosis.

METHODS

Study design Prospective monocentric longitudinal observational study with drug

Population Adults with hATTR amyloidosis with polyneuropathy with a pathogenic TTR mutation (NIS score between 5 and 130 points at baseline) will be enrolled in accordance with the criteria defined in the clinical practice guidelines related to the reference center (FPG).

Inclusion criteria

* Adult patients with hATTR amyloidosis with polyneuropathy with a confirmed TTR disease-causing mutation (NIS score between 5 and 130 points at baseline).
* Patients on hATTR amyloidosis therapy with gene silencers (patisiran or inotersen) and TTR stabilizers (tafamidis at doses of 20 or 61 mg).
* Patients who gave consent to participate in the study.

Exclusion criteria

* Patients aged < 18 years
* Pregnant women
* Patients who refused to give their consent to participate in the study.

Duration of the study The enrolment period in the planned study is 12 months from the date of approval by the local ethics committee. Three visits are scheduled for each patient (baseline; 9 and 18 months). Therefore, the expected participation in the study for each patient will be 18 months. The total duration of the study will be 36 months, of which the last 6 months will be dedicated to data analysis and scientific production.

ENDPOINTS

Primary Endpoint To establish the potential of NfL as a biomarker of severity of polyneuropathy, progression and response to treatment in patients with symptomatic hATTR amyloidosis, in terms of serum NfL levels of patients with hATTR amyloidosis at baseline and after 9 and 18 months of follow-up.

Endpoints secondary Evaluate the correlation between NfL levels and measures of disease severity and progression.

PROCEDURE Demographic and anthropometric data will be collected for all patients at the time of enrollment. In addition, the following evaluations will be carried out.

Plasma NfL levels NfL levels will be measured at baseline, at 9 and 18 months. Serum NfL measurements will be performed with Simple Plex cartridges using Ella equipment (ProteinSimple, San Jose) at Gemelli Polyclinic, the initiator of the study.

Variables

All enrolled patients will undergo the following assessments at each timepoint:

* Stage of familial amyloid polyneuropathy (FAP)
* Polyneuropathy Disability Score (PND)
* neuropathy impairment score (NIS)
* compound autonomic dysfunction test (CADT)
* Questionnaire Norfolk Quality of life-Diabetic neuropathy (Norfolk Qol-DN)
* Cardiological evaluation (echocardiogram and clinical examination)
* Evaluation of dysautonomia (Sudoscan)
* Renal and/or gastrointestinal evaluation (laboratory tests and targeted questions)
* Laboratory tests (NT-proBNP, troponin, creatinine, urinalysis, liver enzymes)

STATISTICAL ANALYSIS PLAN

Sample sizing Since this is a rare disease study for which a limited number of patients per year are observed at the reference center and justified by the primary endpoint of the purely descriptive study, formal sample sizing is not necessary. All subjects belonging to the reference structure will therefore be enrolled within the 12 months foreseen for enrollment. It is estimated in these terms a sample of 40 subjects.

Statistical analysis The sample will be described in its demographic, anthropometric, clinical, instrumental variables, through descriptive statistical techniques. In detail, the qualitative variables will be expressed as absolute frequencies and relative percentages. Quantitative variables, on the other hand, will be reported as mean and standard deviation (SD) or median and interquartile range (IQR), respectively, if they are normally distributed or not. Their distribution will be evaluated in advance by Shapiro Wilk's test. Assessment of the correlation between serum NfL levels at baseline and demographic data (age at onset, age at time of assessment, duration of disease), clinical scales (FAP stage, PND, NIS, NIS-LL score), questionnaires (CADT, Norkfolk QuL-DN) and instrumental evidence (Sudoscan on full and hands, interventricular septal thickness, cardiac markers ) will be carried out through the Spearman or Pearson correlation test, as appropriate. The results will be further graphed in the form of Heatmaps constructed through the R packages "ggpubr" [8], "ggplot2", "ggprism" and "ggsignif" [9-11]. The relationship between NFL levels at 9 and 18 months respectively and the above parameters will be further investigated through a mixed model for repeated measurements (MMRM). The model will include the outcome parameter (NFL) at the end of treatment. Fixed effects will include age at onset and disease duration, follow-up time-points as a categorical variable (baseline, 9 or 18 months), and baseline outcome parameter values. Correlations between repeated measurements will be modeled using a repeating effect with a compound symmetry structure. The models will be rented using the R packages "lme4" and "lmertest" [12,13]. In order to use these models on small samples, a Bartlett-type adjustment will be made by bootstrap resampling with the R package "pbkrtest" [14]. In fact, taking into account that the approximation of the maximum likelihood T-test (LR) statistic to the chi-square distribution in large samples is not accurate on a low scale, the Bartlett correction divides by a correction term, with the adjustment term being an estimate of the first moment of the null distribution of the T-statistic. Statistical significance will be set at a p-value <0.05. All analyses will be performed with R software version 4.2.0 (CRAN ® , R Core, Vienna, Austria, 2022) [15].

Safety/adverse event management Definitions "Adverse event" means any harmful clinical event that occurs in a person who has been given a medicinal product and who does not necessarily have a causal relationship with such treatment.

"Adverse reaction" means the unintended and noxious reaction resulting not only from the authorised use of a medicinal product under normal conditions of use but also from medication errors and uses not in accordance with the indications given in the marketing authorisation, including misuse and abuse of the medicinal product.

"Serious adverse reaction" means an adverse reaction that causes:

* death
* life threatening,
* hospitalization or prolongation of hospitalization,
* severe or permanent invalidity,
* congenital anomalies/birth defects,
* other clinically relevant condition.

Management of adverse events All adverse events will be collected, recorded and evaluated for severity and relationship to investigational and non-investigational medicinal products for the purpose of identifying suspected adverse reactions.

Any suspected adverse reaction will be reported to the National Competent Authority - AIFA, regardless of the severity, according to the post-marketing pharmacovigilance flow, provided for by DM 30 April 2015 and GVP (Good Vigilance Practices) module VI, by communication to the Local Pharmacovigilance Manager for inclusion in the National Pharmacovigilance Network and, where required, to the Ethics Committee.

Suspected adverse drug reactions should be reported to the Local Pharmacovigilance Manager within 48 hours of becoming known, and suspected adverse reactions from biological medicinal products should be reported no later than 36 hours.

STUDY MANAGEMENT Ethical and regulatory considerations This study will be conducted in accordance with the protocol, the Ethical Committee Approval of Policlinico Gemelli, with all applicable regulatory requirements and with the current Good Clinical Practice (GCP) guidelines. GCP adherence publicly ensures the protection of the rights, safety and well-being of trial patients in accordance with the principles of the Helsinki Declaration.

Study documentation, confidentiality and retention All documentation (including personal data) related to the study will be kept as required by local laws and regulations.

The investigator must ensure that the confidentiality of all patients is maintained.

On submitted documents, patients should not be identified by their names, but by numbers or codes assigned to the patient.

End of the study The term of the study is defined by the completion of the last NfL measurement at 18 months for all patients enrolled.

Data quality control and quality assurance Data Management The following patient health information (PHI)/HIPAA identifiers will be collected through a database: name, medical registration numbers, birthdays, gender, race, height, weight, medical and surgical history and dates of diagnoses, laboratory and imaging results, histological findings, drug lists, allergies, clinic, and hospital notes. The information obtained will be limited to the minimum necessary to achieve the purposes of the research study. This study will be monitored by first investigator Dr. Marco Luigetti. The data (name, surname, date of birth) will be coded and stored at the Policlinico Gemelli (Department of Neurology) and will be accessible only to the first researcher and the study group.

Publishing Policy It is understood that after completion of the study, the data should be submitted for publication in a scientific journal and/or for communication at scientific conferences.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hATTR amyloidosis with polyneuropathy with a confirmed TTR disease-causing mutation (NIS score between 5 and 130 points at baseline).
* Patients on hATTR amyloidosis therapy with gene silencers (patisiran or inotersen) and TTR stabilizers (tafamidis at doses of 20 or 61 mg).
* Patients who gave consent to participate in the study.

Exclusion Criteria:

* Patients aged < 18 years
* Pregnant women
* Patients who refused to give their consent to participate in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with hATTR amyloidosis with polyneuropathy with a pathogenic TTR mutation (NIS score between 5 and 130 points at baseline) will be enrolled in accordance with the criteria defined in the clinical practice guidelines related to the reference center (FPG).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in NfL values | 9 and 18 months
  To establish the potential of NfL as a biomarker of severity of polyneuropathy, progression and response to treatment in patients with symptomatic hATTR amyloidosis, in terms of serum NfL levels of patients with hATTR amyloidosis at baseline and after 9 and 18 months of follow-up.and response to treatment in patients with symptomatic in hATTR

SECONDARY OUTCOMES:
NfL levels correlation | 9 and 18 months
  Evaluate the correlation between NfL levels and measures of disease severity and progression.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Luigetti, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, Italy